CLINICAL TRIAL: NCT05732909
Title: The Metabolic Effects of β-hydroxybutyrate on Working Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Diabetes Academy (Other); AP Moeller Foundation (Other); Aarhus University Hospital (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ketomr
Record Dates: First submitted 2023-01-17; First posted 2023-02-17 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2023-01

CONDITIONS: Aging; Metabolism Disorder; Ketonemia; Muscle Disorder
MeSH Terms: conditions — Metabolic Diseases; Ketosis; Muscular Diseases

STUDY DESIGN:
Intervention Model Description: Two-day cross-over design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Ketone, then placebo (Experimental): Ingestion of ketone monoester D-β-hydroxybutyrate / D 1,3 butanediol monoester on first experimental day and ingestion of a fat placebo drink on the second experimental day.
  Interventions: Dietary Supplement: D-β-hydroxybutyrate/D 1,3 butanediol monoester
- First placebo, then ketone (Experimental): Ingestion of a fat placebo drink on the first experimental day followed by ingestion of ketone monoester D-β-hydroxybutyrate / D 1,3 butanediol monoester on the second experimental day.
  Interventions: Dietary Supplement: D-β-hydroxybutyrate/D 1,3 butanediol monoester

INTERVENTIONS:
Dietary Supplement: D-β-hydroxybutyrate/D 1,3 butanediol monoester — Ketone monoester

SUMMARY:
The goal of this clinical trial is to test ketone bodies in healthy elderly and young individuals. The main question it aims to answer are:

• Do ketone bodies improve skeletal muscle function?

Participants will ingest a ketone monoester and skeletal muscle function will then be evaluated by:

* Special magnetic imaging techniques
* Intravenous infusion of tracer-marked nutrients
* Performance tests on a ergometer bike and in a dynamometer

Researchers will compare the outcomes between within the young and elderly groups and between the young and the elderly group to investigate if age has an effect on the outcomes.

DETAILED DESCRIPTION:
BACKGROUND With ageing, skeletal muscles metabolism changes and muscle function declines. This may lead to muscle weakness and increased risk of developing metabolic diseases. Ketone bodies, namely 3-hydroxybutyrate (3-OHB), is an energy substrate that may change the metabolism and improve efficiency of skeletal muscles in a setting of ageing.

OBJECTIVE The study aims to investigate the effects of beta-hydroxybutyrate ingested as a monoester on skeletal muscle function and metabolism during muscle work in young and elderly individuals.

DESIGN Healthy young (20-25 years) and elderly (65-85 years) untrained males will be paired based on age corrected VO2-max. Participants will be evaluated in a double blinded cross-over design on two study days: One day with ketone ester ingestion (D-beta-hydroxybutyrate/D-1,3-butanediol; KetoneAid Pro KE4), one day with ingestion of a volume and calorie and taste matched placebo (lipid emulsion). Blood ketone levels will be kept elevated through a sipping protocol. During both conditions a low glucose dose will be continuously infused to block physiological ketogenesis.

The order of the study days will be randomized and interspaced by at least 4 weeks.

On experimental days, participants meet fasted to perform voluntary contractions with tibialis anterior muscles in a MR compatible dynamometer while oxidative capacity, ATP generation, intramuscular pH, fatiguability and work efficiency is evaluated through 31P-MR spectroscopy.

After, participants will bike at a fixed intensity (~45% of Wmax) while lipid fluxes and glucose oxidation rates are measured by palmitate- and glucose tracer infusions and carbamide-corrected indirect calorimetry over 60 min. This was initially intended for both young and elderly individuals, but only involves the young group, as the elderly group had difficulties completing 60 min cycling.

Lastly on the study days, participants will perform a cycling test as a measure of performance starting at 70 % of Wmax for 5 min thereafter increasing by 10 % of Wmax every 1 min until exhaustion. Muscle biopsies are obtained before (both groups) and just following fixed intensity cycle work (only young group). Adipose tissue biopsies are collected at the beginning of the experimental day (both groups) before ketone/placebo ingestion and after the constant load cycle work (only young group). Blood samples are performed throughout the day to assess substrate levels, hormones and for proteomics analysis.

Before each study day, participant's activity level is measured for 7 days by accelerometry (ActiGraph). Participants will log their diet 3 days prior to each experimental day. Participants are asked to ingest a similar diet 2 days before both experimental days and to withstand from strenuous exercise 2 days prior to both experimental days. Participants are asked not to make any significant changes to their lifestyle while taking part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male 20-25 years old (n = 12) OR male 65-85 years old (n = 12)
* BMI range: 19 to 27
* Stable weight (< 5% change over last 6 months)
* Less than 3 x 60 min of structured exercise per week.

Exclusion Criteria:

* Medication that affect energy metabolism.
* Non-MR-compatible metals or electric devices in the body.
* Anaemia or bleeding disorders.
* Heart, lung or other disease that affects the subjects ability to exercise.
* Smoking.
* Drug abuse.
* Lack of compliance.
* Known allergy towards local anaesthetics.
* Any condition that the principal investigator considers unsuitable for the subject's ability to complete the study.

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Work efficiency | Over 60 minutes on each of the two experimental days.
  External work performed by the ankle during dorsiflexion per ATP consumed. ATP consumption is assessed by 31P-MRS while external force is measured by the dynamometer.

SECONDARY OUTCOMES:
Oxidative capacity | Over 20 minutes at each of the two experimental days.
  Assessed by 31P-MRS as phosphocreatine resynthesis.
Glucose oxidation rates (only young group) | At 10 minute intervals over the last 30 min of the 90 min fixed intensity cycling on each experimental day.
  Assessed by measuring tracer dilution from blood samples obtained during 3H-glucose infusion while cycling at a fixed intensity.
Palmitate flux (only young group) | At 10 minute intervals over the last 30 min of the 90 min fixed intensity cycling on each experimental day.
  Assessed by measuring tracer dilution from blood samples obtained during 3H-palmitate infusion while cycling at a fixed intensity.
ATP generation | Over 30 minutes at each of the two experimental days.
  ATP generated from different pathways (glycolytic, oxidative, phosphocreatine) assessed by 31P-MRS.
Mitochondrial function | Just before and immediately after the constant load cycling at each of the two experimental days.
  Assessed by high-resolution respirometry on muscle biopsies
Intramuscular pH | Over 60 minutes at each of the two experimental days.
  Measurements at rest rest and during work assessed by 31P-MRS
Blood 3-OHB | During each of the two experimental days
  Blood concentration measured by blood sampling
Blood glucose | During each of the two experimental days
  Blood concentration measured by blood sampling
Blood free fatty acids | During each of the two experimental days
  Blood concentration measured by blood sampling
Cycle performance | 5-8 minutes during each of the two experimental days
  Assessed by a performance test on a bike ergometer with incremental load. The test continues until failure. The test outcome is the power generated at time of failure.
Rating of perceived exertion (only young group) | After 30, 60 and 90 minutes of fixed intensity cycling and just after the incremental performance test.
  Subjective measure of exertion during cycling evaluated by reporting on a number assessment scale (Borg scale (6-20)).
Tibialis anterior fatigue | Over 3 minutes on each of the two experimental days.
  Tibialis anterior fatigue assessed by the dynamometer during 3 minutes of dorsiflexion at a fixed resistance.
Blood growth hormone | During experimental days
  Blood concentration measured by blood sampling
Blood insulin | During each of the two experimental days
  Blood concentration measured by blood sampling
AMPK phosphorylation (only young group) | Just before and immediately after the constant load cycling at each of the two experimental days.
  From muscle biopsies
Blood glucagon | During each of the two experimental days
  Blood concentration measured by blood sampling
Blood pH | During each of the two experimental days
  Assessed from arterial blood samples
Blood catecholamines | During each of the two experimental days
  Blood concentration measured by blood sampling
Blood cortisol | During each of the two experimental days
  Blood concentration measured by blood sampling
Intramuscular lipid content | At the beginning and at the end of each of the two experimental days
  Concentration measured in muscle biopsies
Intramuscular glycogen content | Just before and immediately after the constant load cycling at each of the two experimental days.
  Concentration measured in muscle biopsies

OTHER OUTCOMES:
Blood haemoglobin | Measured at the beginning and the end of each experimental day
  Blood concentration measured by blood sampling
Blood Sodium | Measured at the beginning and the end of each experimental day
  Blood concentration measured by blood sampling
Blood potassium | Measured at the beginning and the end of each experimental day
  Blood concentration measured by blood sampling
Blood creatinine | During each of the two experimental days
  Blood concentration measured by blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Niels Jessen, Professor, Study Director — Aarhus University Hospital
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus, Aarhus N, Denmark

REFERENCES:
- [Derived] Andersen OE, Larsen RG, Moller N, Stouge A, Ringgaard S, Overgaard K, Jessen N. Ketone Monoester Increases Skeletal Muscle Power and Energy Turnover in Older but Not Young Men Without Affecting Metabolic Economy: A Controlled, Double Blind, Cross-Over Trial. Acta Physiol (Oxf). 2026 Mar;242(3):e70161. doi: 10.1111/apha.70161. PMID 41644499